CLINICAL TRIAL: NCT04369833
Title: Development of Continuous Glucose Monitoring System Cohort for Personalized Diabetes Prevention and Management Platform Based on Artificial Intelligence Model Using Mathematical Analysis
Brief Title: Development of Continuous Glucose Monitoring System Cohort for Personalized Diabetes Prevention and Management Platform
Status: Completed | Type: Observational
Sponsor: Pusan National University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: H-2003-033-088
Record Dates: First submitted 2020-04-27; First posted 2020-04-30 (Actual); Results first posted 2022-05-09 (Actual); Last update posted 2022-05-09 (Actual); Status verified 2022-02

CONDITIONS: PreDiabetes; Glucose Metabolism Disorders; Diabetes Mellitus
MeSH Terms: conditions — Prediabetic State; Glucose Metabolism Disorders; Diabetes Mellitus | interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Biospecimen Retention: Samples Without DNA — blood sample (for HbA1c, Total cholesterol, LDL-C, HDL-C, Triglyceride, aspartate aminotransferase, alanine aminotransferase, Creatinine, free fatty acid etc), Feces (for evaluating microbiomes)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- continuous glucose monitoring group: all participants wearing a continuous glucose monitoring device
  Interventions: Device: continuous glucose monitoring system

INTERVENTIONS:
Device: continuous glucose monitoring system — wearing continuous glucose monitoring device (iPro2 professional continuous glucose monitoring, MedtronicⓇ, California, USA)

SUMMARY:
The purpose of this study is to collect a variety of clinical data and blood glucose changes using a continuous glucose monitoring device for high-risk diabetes patients (prediabetes) in order to develop a personalized diabetes prevention and management platform based on artificial intelligence model using mathematical analysis.

DETAILED DESCRIPTION:
After being informed about the study and potential risks, all patients giving written informed consent wear a continuous glucose monitoring device ("iPro2" professional continuous glucose monitoring, MedtronicⓇ, California, USA) and smart band ("Fitbit Inspire HR", FitbitⓇ, California, USA) for 1 week.

During this period, all patients are tested oral glucose tolerance test and take a standard diet (calorie calculated) at morning.

The patient's data from this study is compared to a predicted values by mathematical analysis model for diabetes prevention.

ELIGIBILITY:
Inclusion Criteria:

* Above 18 years old.
* Prediabetes

  1. Fasting plasma glucose : 100~125mg/dL, fasting is defined as no caloric intake for at least 8 hours.

     OR
  2. 2-hour plasma glucose during 75g oral glucose tolerance test : 140 ~ 199mg/dL

     OR
  3. Glycated hemoglobin(HbA1c) : 5.7~6.4% (39-47mmol/mol)

Exclusion Criteria:

* with a history of newly diagnosed and treated cancer within the last 5 years
* with a history of hospitalization for active disease within the last 3 months
* with a history of severe cardiovascular disease within the last 3 months
* with a history of steroid treatment in the last 3 months
* people who have had major surgery planned within the last 3 months or who have had surgery within 3 months
* people who are pregnant or have been in the last 3 months after giving birth

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects of pre-diabetes who visited the Department of Internal Medicine and division of Endodrinology & Metabolism and the Health Examination Center, Pusan National University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2020-05-11 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sang soo Kim, Master, Principal Investigator — Pusan National University Hospital
Locations (1):
- Pusan national university hospital, Busan, South Korea

IPD SHARING:
Plan to Share IPD: No
The data are not publicly available due to privacy or ethical restrictions.

REFERENCES:
- [Background] Kang H, Han K, Jo J, Kim J, Choi MY. Systems of pancreatic beta-cells and glucose regulation. Front Biosci. 2008 May 1;13:6421-31. doi: 10.2741/3163. PMID 18508669
- [Background] Hansen BC, Jen KC, Belbez Pek S, Wolfe RA. Rapid oscillations in plasma insulin, glucagon, and glucose in obese and normal weight humans. J Clin Endocrinol Metab. 1982 Apr;54(4):785-92. doi: 10.1210/jcem-54-4-785. PMID 7037815
- [Background] Lang DA, Matthews DR, Peto J, Turner RC. Cyclic oscillations of basal plasma glucose and insulin concentrations in human beings. N Engl J Med. 1979 Nov 8;301(19):1023-7. doi: 10.1056/NEJM197911083011903. PMID 386121
- [Background] Mendes-Soares H, Raveh-Sadka T, Azulay S, Edens K, Ben-Shlomo Y, Cohen Y, Ofek T, Bachrach D, Stevens J, Colibaseanu D, Segal L, Kashyap P, Nelson H. Assessment of a Personalized Approach to Predicting Postprandial Glycemic Responses to Food Among Individuals Without Diabetes. JAMA Netw Open. 2019 Feb 1;2(2):e188102. doi: 10.1001/jamanetworkopen.2018.8102. PMID 30735238
- [Background] Kim BY, Won JC, Lee JH, Kim HS, Park JH, Ha KH, Won KC, Kim DJ, Park KS. Diabetes Fact Sheets in Korea, 2018: An Appraisal of Current Status. Diabetes Metab J. 2019 Aug;43(4):487-494. doi: 10.4093/dmj.2019.0067. Epub 2019 Jul 17. PMID 31339012
- [Background] Ha KH, Lee YH, Song SO, Lee JW, Kim DW, Cho KH, Kim DJ. Development and Validation of the Korean Diabetes Risk Score: A 10-Year National Cohort Study. Diabetes Metab J. 2018 Oct;42(5):402-414. doi: 10.4093/dmj.2018.0014. Epub 2018 Jul 6. PMID 30113144
- [Background] Lee YH, Bang H, Kim HC, Kim HM, Park SW, Kim DJ. A simple screening score for diabetes for the Korean population: development, validation, and comparison with other scores. Diabetes Care. 2012 Aug;35(8):1723-30. doi: 10.2337/dc11-2347. Epub 2012 Jun 11. PMID 22688547
- [Background] Zeevi D, Korem T, Zmora N, Israeli D, Rothschild D, Weinberger A, Ben-Yacov O, Lador D, Avnit-Sagi T, Lotan-Pompan M, Suez J, Mahdi JA, Matot E, Malka G, Kosower N, Rein M, Zilberman-Schapira G, Dohnalova L, Pevsner-Fischer M, Bikovsky R, Halpern Z, Elinav E, Segal E. Personalized Nutrition by Prediction of Glycemic Responses. Cell. 2015 Nov 19;163(5):1079-1094. doi: 10.1016/j.cell.2015.11.001. PMID 26590418
- [Background] Shapiro ET, Tillil H, Polonsky KS, Fang VS, Rubenstein AH, Van Cauter E. Oscillations in insulin secretion during constant glucose infusion in normal man: relationship to changes in plasma glucose. J Clin Endocrinol Metab. 1988 Aug;67(2):307-14. doi: 10.1210/jcem-67-2-307. PMID 3292558
- [Background] Kraegen EW, Young JD, George EP, Lazarus L. Oscillations in blood glucose and insulin after oral glucose. Horm Metab Res. 1972 Nov;4(6):409-13. doi: 10.1055/s-0028-1094019. No abstract available. PMID 4655495
- [Background] Simon C, Brandenberger G, Follenius M. Ultradian oscillations of plasma glucose, insulin, and C-peptide in man during continuous enteral nutrition. J Clin Endocrinol Metab. 1987 Apr;64(4):669-74. doi: 10.1210/jcem-64-4-669. PMID 3102544

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Continuous Glucose Monitoring Group
Started | 130
Completed | 129
Not Completed | 1

BASELINE CHARACTERISTICS:
Population: Patients who have high risk for developing diabetes with wearing CGM.
Arm/Group | Continuous Glucose Monitoring Group
Number analyzed (Participants) | 129
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.6 (12.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 96
  Male | 33
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 129
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  South Korea | 129
Mean CGM glucose [Mean (Standard Deviation); unit: mg/dL] | 122.6 (15.5)
the coefficient of variation of CGM glucose [Mean (Standard Deviation); unit: percentage of coefficient of variation] | 19.6 (6.4)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Insulin Resistance
Description: the prevalence of insulin resistance in participants was measured. Insulin resistance was calculated by HOMA-IR(homeostatic model assessment of insulin resistance), QUICKI (quantitative insulin sensitivity check index) and Matsuda index
Time Frame: 1 week
Measure: Count of Participants; unit: Participants
Arm/Group | Continuous Glucose Monitoring Group
Number analyzed (Participants) | 129
Participants | 69

ADVERSE EVENTS:
Time Frame: 1 week
Arm/Group | Continuous Glucose Monitoring Group
All-Cause Mortality (participants affected / at risk) | 0/129
Serious Adverse Events (participants affected / at risk) | 0/129
Other Adverse Events (participants affected / at risk) | 1/129
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Continuous Glucose Monitoring Group (N=129)
bleeding on CGM insertion site (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-15): https://cdn.clinicaltrials.gov/large-docs/33/NCT04369833/Prot_SAP_000.pdf